CLINICAL TRIAL: NCT01801904
Title: A Phase 2 Study of Panitumumab in Patients With Cetuximab-refractory Metastatic Colorectal Cancer
Acronym: PACER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Collaborators: Azienda Ospedaliera G. Rummo (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PACER; 2010-024490-39 (EudraCT Number)
Record Dates: First submitted 2013-01-15; First posted 2013-03-01 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: cetuximab-refractory
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab (Experimental)
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — 6mg/kg IV given every 2 weeks until disease progression or unacceptable toxicity

SUMMARY:
The purpose of this study is to assess if panitumumab is active enough to warrant comparative studies in patients with metastatic colorectal cancer that has progressed after treatment with cetuximab.

DETAILED DESCRIPTION:
The study was amended with modification of inclusion criteria (from wild-type tumor KRAS gene to wild-type RAS gene, including KRAS and NRAS exons 2, 3 and 4)

RAS mutational status of tumors of patients enrolled before amendment 1 approval will be centrally revised. Patients whose tumors will result RAS mutated at the biomarkers central revision, will be replaced. Therefore, the overall sample size at both the stages may be higher than the one initially planned.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of metastatic colorectal adenocarcinoma
* a wild-type RAS tumor (mutational status has to be determined by an experienced laboratory using validated test methods for detection of KRAS exons 2, 3, and 4, and NRAS exons 2, 3, and 4
* Failure from previous treatment with fluoropyrimidine, oxaliplatin and irinotecan. Patients may or may not have been treated with bevacizumab.
* Documented disease progression following a treatment with cetuximab in patients who showed either an objective response after 8 weeks or stable disease after 16 weeks of cetuximab treatment.
* Age at least 18 years
* ECOG Performance Status 0-2
* Neutrophils at least 1,500 mm3, platelets at least 100,000 mm3, and hemoglobin at least 9 g/dL
* Bilirubin level less than 1.5 times ULN
* AST (SGOT) and ALT (SGPT) not greater than 2.5 times ULN (or 5 times ULN in presence of liver metastasis)
* Serum creatinine less than 1.5 times ULN
* Effective contraception, if the risk of conception exists
* Life expectancy at least 3 months
* Written informed consent

Exclusion Criteria:

* Symptomatic brain metastasis
* Interstitial pneumonitis or pulmonary fibrosis
* Any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or non melanoma skin cancer)
* Chemotherapy, radiotherapy or immunotherapy within the past 4 weeks
* Any unstable systemic disease (including active infections, any significant hepatic, renal or metabolic disease), metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of study drugs or render the patient at high risk from treatment complications
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-12; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
number of patients alive and without disease progression | 2 months
  progression of disease within 2 months from registration according to RECIST criteria, and death for any cause within 2 months from registration

SECONDARY OUTCOMES:
response rate | up to 40 weeks
  Response assessed per patients at weeks 8,16,24,32,40 and every 3 months thereafter, using RECIST criteria
progression free survival | 9 months
overall survival | one year
worst grade toxicity per patient | every 2 weeks for up to 6 months
  worst grade toxicity (according to Common Terminology Criteria for Adverse Events version 3) per patient

OTHER OUTCOMES:
gene expression on tumor tissue | one year
  exploratory analysis of tumor-tissue for biological or genomic determinants of outcome of BRAF and P13K mutation status, EGFR and PTEN expression status

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Daniele, M.D., Principal Investigator — Azienda Sanitaria Rummo, Benevento, Division of Medical Oncology; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute Naples, Italy; Director Clinical Trials Unit; Ciro Gallo, M.D., Ph.D, Principal Investigator — Second University of Naples, Italy; Chair of Medical Statistics; Antonio Gasbarrini, M.D., Principal Investigator — Università Cattolica del S. Cuore, Policlinico Gemelli, Roma; Giacomo Carteni', M.D., Principal Investigator — Ospedale Antonio Cardarelli, Napoli
Locations (5):
- Italy (5):
  - Azienda Ospedaliera G. Rummo, Benevento, BN
  - Ospedale Fatebenefratelli, Benevento
  - A.O.U. Policlinico Federico II, Napoli
  - Istituto Nazionale dei Tumori, Napoli
  - Casa Sollievo Sofferenza, S. Giovanni Rotondo

REFERENCES:
- [Derived] Piccirillo MC, Avallone A, Carlomagno C, Maiello E, Rosati G, Alabiso O, Nasti G, De Placido S, Latiano TP, Bilancia D, Ottaiano A, De Stefano A, Romano C, Silvestro L, Nappi A, Cassata A, Giordano P, Iaffaioli RV, Normanno N, Perrone F, Daniele B. Multicenter Single-Arm, Two-Stage Phase 2 Study of Panitumumab in Patients With Cetuximab-Refractory Metastatic Colorectal Cancer: The PACER Trial. Clin Colorectal Cancer. 2020 Dec;19(4):270-276. doi: 10.1016/j.clcc.2020.05.009. Epub 2020 May 29. PMID 32631788